CLINICAL TRIAL: NCT04196348
Title: Characterization of Intestinal Hormone and Glucose Dynamics to Unravel the Antidiabetic Effect of Bariatric Surgery
Brief Title: Surgical Innovation for Diabetes Treatment
Acronym: SURIDIAB-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Sao Sebastiao (Other)
Collaborators: Instituto de Ciências Biomédicas Abel Salazar (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Marta Guimarães, SURIDIAB-1 Principal investigator, Hospital de Sao Sebastiao
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hsebastião
Record Dates: First submitted 2019-05-10; First posted 2019-12-12 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: Bariatric Surgery; Gastric Bypass; Obesity; Type 2 Diabetes Mellitus; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short BPL RYGB in glucose-tolerant participants (Active Comparator): Procedure: short biliopancreatic limb (BPL) Roux en Y Gastric Bypass (RYGB) Obese patients without type 2 diabetes mellitus (T2DM) to be submitted to short BPL (n=10)
  Interventions: Procedure: Short BPL RYGB
- Long BPL RYGB in glucose-tolerant participants (Active Comparator): Procedure: long BPL RYGB Obese patients with metabolic syndrome without T2DM to be submitted to long BPL (n=10)
  Interventions: Procedure: Long BPL RYGB
- Long BPL RYGB in diabetic participants (Active Comparator): Procedure: long BPL RYGB Obese patients with metabolic syndrome and T2DM to be submitted to long BPL (n=10)
  Interventions: Procedure: Long BPL RYGB

INTERVENTIONS:
Procedure: Short BPL RYGB — Alimentary limb (AL) with 120 cm and BPL with 100 cm.
  Arms: Short BPL RYGB in glucose-tolerant participants
Procedure: Long BPL RYGB — AL with 120 cm and BPL with 200 cm.
  Arms: Long BPL RYGB in diabetic participants; Long BPL RYGB in glucose-tolerant participants

SUMMARY:
This study will determine how two variants of gastric bypass induce changes in dynamic endocrine response in the fasting and post-prandial state, both before and at different time points after the surgical interventions.

This study will monitor the endocrine dynamics after different anatomical modifications produced by Roux-en-Y gastric bypass procedures in diabetic participants and normoglycemic participants, to gain insights into the mechanisms beyond the metabolic improvement after the two surgical variants through participants re-evaluation at different time points.

DETAILED DESCRIPTION:
Abstract

Obesity prevalence is a major risk factor for the onset of type 2 diabetes. Diabetic patients are frequently overweight or obese and diabetes complications are the main cause of obesity-related morbimortality, demanding proper and effective clinical management.

Bariatric surgery, originally conceived for obesity treatment, has proven not only to be the most effective weight loss intervention but also for comorbidity management, with a strong impact on type 2 diabetes. As the antidiabetic effects of bariatric surgery largely exceed the metabolic improvement predicted by the caloric restriction and weight loss, which are mostly driven by the enteroendocrine response, this challenges the academic and medical communities with the need to learn how to leverage the enteroendocrine system to achieve glucose homeostasis.

Supported on the investigators' previous work focusing on gastro-intestinal hormones and glucose metabolism after bariatric surgery, the investigators now aim to monitor the intestinal hormone after different anatomical modifications produced by Roux-en-Y gastric bypass procedures in diabetic participants and normoglycemic individuals. The utmost goal will be to unravel the endocrine mechanisms beyond the metabolic improvement observed after the surgical manipulations, towards the identification of novel targets for hormone based treatments in an individualised clinical approach.

Study Overview: Participants in this study will be submitted to either short or long BPL RYGB surgery. Participants visits will be scheduled before surgery and after surgery at 3, 6 and 12 months for detailed participants assessment that will include anthropometric and biochemical evaluation and the performance of a MMTT with plasma sampling for hormonal profiles.

Participant Enrolment: Participants will be selected from the cohort of patients referred for multidisciplinary evaluation by the clinical team for surgical treatment of obesity of the Centro Hospitalar Entre Douro e Vouga (CHEDV). Participants found to be suitable according to the entry criteria and accept to participate will be enrolled in the study and assigned to one of the three study groups according to participants clinical features.

Study Chair: Mário Nora, MD

Principal Investigator: Marta Guimarães, MD, PhD

ELIGIBILITY:
Inclusion Criteria:

* BMI between 35 and 45 kg/m2 with indication for bariatric surgery
* Aged between 18 and 65 years at surgery

Exclusion Criteria:

* Unwillingness, inability or intolerance to complete the MMTT (ingest 200 mL in 15 minutes or less)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Body mass index (BMI) combines height (in meters) and weight (in kilograms) and is calculated as weight over (height)^2. Therefore, it will be reported in kg/m^2. This parameter will be determined at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) at presential visits to the clinic.
Change in glycated haemoglobin | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glycated haemoglobin (HbA1c) will be measured in percentage (%). This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post- surgery) through routine complete biochemical evaluation.
Change in glucose dynamic profile | Time Frame: From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glucose will be measured in mmol/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in insulin dynamic profile | Time Frame: From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Insulin will be measured in mIU/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in glucagon dynamic profile | Time Frame: From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glucagon will be measured in pmol/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in GLP-1 dynamic profile | Time Frame: From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glucagon-like peptide-1 (GLP-1) will be measured in pmol/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in GIP dynamic profile | Time Frame: From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glucose-dependent insulinotropic polypeptide (GIP) will be measured in pmol/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- São Sebastião Hospital, Santa Maria da Feira, Aveiro District, Portugal

IPD SHARING:
Plan to Share IPD: No